CLINICAL TRIAL: NCT06050616
Title: Multimodal Longitudinal and Machine Learning-based Predictive Modelling to Understand the Development of Eating Disorders
Brief Title: Multimodal Longitudinal and Predictive Modelling to Understand Eating Disorder Development
Acronym: ESTRA-BED
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Delosis Limited (Unknown); NeuroSpin (Unknown)
Responsible Party: Principal Investigator, Zuo Zhang, Principal Investigator, King's College London
Other Study IDs: IRAS326571; MRF-058-0014-F-ZHAN-C0866 (Other Grant/Funding Number: Medical Research Foundation, UK); 23/NW/0232 (Other: NorthWest-Greater Manchester South Research Ethics Committee)
Record Dates: First submitted 2023-09-06; First posted 2023-09-22 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Binge-Eating Disorder; Anorexia Nervosa; Bulimia Nervosa
Keywords: Eating Disorders; Binge-Eating Disorder; Anorexia Nervosa; Bulimia Nervosa; Neuroimaging
MeSH Terms: conditions — Binge-Eating Disorder; Anorexia Nervosa; Bulimia Nervosa; Feeding and Eating Disorders | interventions — Magnetic Resonance Spectroscopy; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Two EDTA tubes and 2 Tempus tubes of blood will be collected. A urine sample (stored in 2 x 10ml tubes) will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- binge eating disorder: Participants with a current binge eating disorder, as assessed by the Eating Disorder Diagnostic Screen (DSM-5 version). These participants have been recruited as part of the STRATIFY study. An additional 30 participants will be recruited in this study to enlarge the sample size, using the same study procedure and assessments in the STRATIFY study.
  Interventions: Other: MRI scans; Other: Psychological measures; Other: Life experiences; Biological: Blood and urine samples; Other: Mental health symptoms
- anorexia nervosa: Participants with current anorexia nervosa, as assessed by the Eating Disorder Diagnostic Screen (DSM-5 version).. These participants have been recruited as part of the STRATIFY study. Their data will be used in this study.
  Interventions: Other: MRI scans; Other: Psychological measures; Other: Life experiences; Biological: Blood and urine samples; Other: Mental health symptoms
- bulimia nervosa: Participants with current bulimia nervosa, as assessed by the Eating Disorder Diagnostic Screen (DSM-5 version). These participants have been recruited as part of the STRATIFY study. Their data will be used in this study.
  Interventions: Other: MRI scans; Other: Psychological measures; Other: Life experiences; Biological: Blood and urine samples; Other: Mental health symptoms
- healthy controls: Healthy controls are selected from the IMAGEN study at the third follow-up (~age 22 years) who do not exhibit any psychiatric disorder. Their data will be used in this study. IMAGEN and STRATIFY are sister studies that employ matched study protocols.
  Interventions: Other: MRI scans; Other: Psychological measures; Other: Life experiences; Biological: Blood and urine samples; Other: Mental health symptoms

INTERVENTIONS:
Other: MRI scans — Neuroimaging data will be collected with magnetic resonance imaging (MRI).
  Structural neuroimaging will include T1 and T2-weighted scans, and diffusion tensor imaging (DTI).
  Functional neuroimaging will include scans under the stop-signal task, monetary incentive delay task, and emotional faces task, and resting state.
Other: Psychological measures — Cognitive performance assessed by Wechsler Adult Intelligence Scale 4th Edition.
  Personalities assessed by NEO Five-Factor Inventory (NEO-FFI), Substance Use Risk Profile Scale (SURPS), and Temperament and Character Inventory (TCI).
  Other psychological assessments include Interpersonal Reactivity Index, Perceived Stress Scale, Kirby Monetary Choice Questionnaire, Passive Avoidance Learning Paradigm, and Stimulus-response compatibility.
Other: Life experiences — Self-report questionnaires on experiences of bullying and trauma.
Biological: Blood and urine samples — Blood and urine samples will be collected but will not undergo analysis in this study. Instead, these samples will be stored in a biobank for potential analysis in future research.
Other: Mental health symptoms — Symptoms of depression measured by the Patient Health Questionnaire -8.
  Symptoms of generalised anxiety, obsessives compulsive disorder, attention deficit hyperactivity disorder, social phobia, specific phobia, agoraphobia, post-traumatic stress disorder, measured by the Development and Well-Being Assessment (DAWBA).
  Harmful drinking measured by the Alcohol use disorders identification test.
  Drug use measured by the European School Survey Project on Alcohol and Other Drugs (ESPAD).
  Suicide risk measured by the the Mini International Neuropsychiatric Interview.

SUMMARY:
The aim of this observational study is to elucidate the biopsychosocial (including neural, psychological, and social) basis of eating disorders (EDs).

The investigators will use functional and structural neuroimaging, psychological as well as environmental data to identify both shared and distinct behavioural/neural processes across ED diagnoses. The investigators will use advanced statistical methods such as machine learning based models.

The investigators will carry out analysis on the data already collected in the STRATIFY (Brain network based stratification of reinforcement-related disorders, IRAS ID 218030) and IMAGEN studies (Reinforcement-related behaviour in normal brain function and psychopathology, reference PNM/10/11-126), including participants with Anorexia Nervosa (N=60), Bulimia Nervosa (N=52), Binge eating disorder (N=27) and healthy controls. In addition, the investigators will recruit 30 new participants with a binge eating disorder using the original STRATIFY study protocol to enlarge the binge eating disorder group, so that its sample size is comparable to the other groups.

Participants will complete online questionnaires, take an online clinical interview, and undergo a research visit, including brain scans, collection of blood and urine samples, and assessment using a range of cognitive and behavioural measures.

DETAILED DESCRIPTION:
Eating disorders (EDs) are serious mental illnesses that involve a range of disturbed emotions, cognitions, and behaviours related to body shape/weight and eating. The causes of EDs are complex and involve many biological, psychological, and social factors. The investigators are interested in understanding the connections between a range of biological, psychological, social factors and eating disorders. This will help us understand the basis of diagnostic classifications, which will promote early intervention and the identification of new areas to target in treatments.

The investigators will analyse the data already collected in the STRATIFY (Brain network based stratification of reinforcement-related disorders, IRAS ID 218030) and IMAGEN studies (Reinforcement-related behaviour in normal brain function and psychopathology, reference PNM/10/11-126), including patients with Anorexia Nervosa (N=60), Bulimia Nervosa (N=52), Binge eating disorder (N=27) and healthy controls. In addition, the investigators will recruit 30 new participants with a current binge eating disorder using the original STRATIFY protocol to enlarge the binge eating disorder group, so that its sample size is comparable to the other groups. Due to funding limitations, 18 participants will take part in the full assessments, including the research visit (MRI scans, blood, and urine samples). The other 12 participants will take part in the online parts of the assessments only, without the research visit.

The investigators will use neuroimaging, cognitive, psychological and life events data to assess if behavioural/neural processes differentiate one eating disorder from another and if there are similar processes across ED diagnoses. The investigators will use advanced statistical methods such as machine learning based models.

The investigators will further test whether the identified behavioural and neurological processes can predict future disease risk, by using data from the IMAGEN study - a longitudinal population-based genetic and imaging study - that involves over 2000 participants followed up from adolescence to early adulthood.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers, all ethnicities.
* Age of 18 to 30.
* Sufficient in English (due to validity of neuropsychological measures).
* current DSM-5 binge eating disorder.

Exclusion Criteria:

* People with brain injuries including stroke, tumours, epilepsy, neurodegenerative or other neurological disorders.
* People who are deaf or have significant hearing problems or a hearing aid that cannot be removed.
* People who are blind or have significant vision difficulties (correct near vision of 20/100 or worse in both eyes).
* People with type I or type II diabetes.
* People who are heavily medicated for serious illness (other than for mental illness).
* People who are pregnant or any possibility of being pregnant.
* People with restricted mobility, including inability to lie flat for 1.5 hours.
* People who have a history of anorexia nervosa and have not restored their body weight in the past 6 months.
* People who have participated in the STRATIFY, ESTRA or IMAGEN studies previously.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will be recruited via online and physical posters among people living in or near London, UK, and from eating disorder clinics in London.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
Eating disorder diagnosis | Administered at the screening phase and within two weeks of the other assessments.
  The Eating Disorder Diagnostic Scale (DSM-5 version) will be used to assess whether the participants meet the diagnostic criteria of anorexia nervosa, bulimia nervosa, or binge eating disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Zuo Zhang, PhD, Principal Investigator — King's College London
Locations (1):
- Institute of Psychiatry, Psychology & Neuroscience, King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data are to be shared. Data will be pseudonymised before sharing.
Supporting Information: Study Protocol
Time Frame: starting 6 months after publication of the research findings
Access Criteria: A short data access application must be submitted to the principle investigator, including specific research questions, choice of variables, and plans for analysis and publication. The principle investigator will discuss with the STRATIFY Executive Committee (chaired by the Centre for Population Neuroscience and Stratified Medicine, Charité - Universitätsmedizin Berlin) about the application, and inform the applicant of the outcome.